CLINICAL TRIAL: NCT03604380
Title: STATE Trial: SusTained Attention Training to Enhance Sleep (Phase I- Remote Trial Arm)
Brief Title: STATE Trial: SusTained Attention Training to Enhance Sleep - Remote
Acronym: STATE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Posit Science Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PSC-0510-18
Record Dates: First submitted 2018-07-11; First posted 2018-07-27 (Actual); Last update posted 2020-12-02 (Actual); Status verified 2020-11

CONDITIONS: Insomnia Chronic
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Treatment (Experimental): Computerized plasticity-based adaptive cognitive training requiring a total maximum of 36 treatment sessions, up to 7 sessions per week, 36 minutes per session.
  Interventions: Other: Computerized Plasticity-Based Adaptive Cognitive Training
- Active Comparator (Active Comparator): Commercially available computerized training requiring a total maximum of 36 treatment sessions, up to 7 sessions per week, 36 minutes per session.
  Interventions: Other: Active Comparator

INTERVENTIONS:
Other: Computerized Plasticity-Based Adaptive Cognitive Training — Computerized plasticity-based adaptive cognitive training requiring a total maximum of 36 treatment sessions, up to 7 sessions per week, 36 minutes per session.
  Arms: Experimental Treatment
Other: Active Comparator — Commercially available computerized training requiring a total maximum of 36 treatment sessions, up to 7 sessions per week, 36 minutes per session.
  Arms: Active Comparator

SUMMARY:
This study is a validation study to document the acceptability of the Tonic and Phasic Alertness Training (TAPAT) program in older adults with chronic late-life insomnia. The goal of this study is to employ a computerized attention-training program, TAPAT, designed for chronic late-life insomnia in a remote, randomized, controlled trial to assess feasibility and initial efficacy in this population.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be 55 years of age or older.
* Participant must meet criteria for clinical insomnia - moderate severity based on the Insomnia Severity Index.
* Participant must be a fluent English speaker.
* Participant must have adequate visual, auditory, and motor capacity to use computerized intervention.
* Participant must have a computer and access to the Internet.

Exclusion Criteria:

* Participants with untreated psychiatric conditions, including substance abuse/dependence disorders, untreated obstructive sleep apnea, diagnosis of other sleep disorders (e.g., restless legs syndrome), recent hospitalization, ongoing chemotherapy or other cancer treatment, and concurrent engagement in another insomnia treatment.
* Participants enrolled in another concurrent research study.
* Participants using computer-based cognitive training programs or has used them within a month of the consent date.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2018-07-10 (Actual); Primary Completion 2020-11-04 (Actual); Study Completion 2020-11-04 (Actual)

PRIMARY OUTCOMES:
Sleep efficiency scores on the Pittsburg Sleep Quality Index | 6 months
Sleep duration scores on the Pittsburg Sleep Quality Index | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Van Vleet, PhD, Principal Investigator — Posit Science Corporation
Locations (1):
- Posit Science Corporation, San Francisco, California, United States